CLINICAL TRIAL: NCT01546974
Title: Prospective Analysis of the Incidence of Ventilator-associated Pneumonia Related to the Humidification System: Heat and Moisture Exchanger Versus Heated Humidification
Brief Title: Ventilator-associated Pneumonia (VAP) and Humidification System
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, Coordinator ICU, Hospital Sao Domingos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: hsd2012; CEP026/2011 (Other: Hospital Sao Domingos)
Record Dates: First submitted 2012-03-03; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-01

CONDITIONS: Ventilator-associated Pneumonia
Keywords: Mechanical Ventilation; Humidification system; Patients submitted to mechanical ventilation for at least 48 hours
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HME filter (Experimental)
  Interventions: Device: HME filter Twin Star 55, Drager Medical, Germany
- Heated humidificator MR 730 Fisher & Paykel (Experimental)
  Interventions: Device: Heated humidification

INTERVENTIONS:
Device: HME filter Twin Star 55, Drager Medical, Germany
  Arms: HME filter
Device: Heated humidification
  Arms: Heated humidificator MR 730 Fisher & Paykel

SUMMARY:
The purpose of this study is to determine which humidification system is more effective in preventing pneumonia in mechanically ventilated patients. The study will compare a heat and moisture exchanger versus heated humidification.

ELIGIBILITY:
Inclusion Criteria:

* Patients expected to require mechanical ventilation for at least 48 hours

Exclusion Criteria:

* Patients < 18 yo and pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
VAP incidence

SECONDARY OUTCOMES:
Duration of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: JOSE R AZEVEDO, MD, Study Chair — Director ICU
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil